CLINICAL TRIAL: NCT04376918
Title: Evaluating the Safety and Efficacy of the Bag-Valve-Guedel Adaptor in Anesthetized Bearded Men in Comparison to the Standard Face Mask - a Prospective, Randomized Cross-over Clinical Trial
Brief Title: Bag-Valve-Guedel Adaptor Vs Common Face Mask for the Ventilation of Anesthetized Bearded Men
Acronym: BVGA02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Lilach Gavish, Study Director, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0172-20-HMO
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ventilation
Keywords: ventilation; airway management; intubation; emergency responders
MeSH Terms: conditions — Respiratory Aspiration | interventions — Masks

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (sequence randomization), controlled (cross over)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Begin with BVGA (Active Comparator): After initial anesthesia induction, anesthetized volunteers will be ventilated through through the BVGA for 2 minutes and then through the face-mask for 2 minutes. The normal anesthesia procedures will then be resumed.
  The BVGA enables the direct connection of a bag valve device to a Guedel, eliminating the need for a face mask during ventilation The Mask is a classic face mask
  Interventions: Device: Begin with BVGA
- Begin with Face-mask (Active Comparator): After initial anesthesia induction, anesthetized volunteers will be ventilated through the face mask for 2 minutes and then through the BVGA for 2 minutes. The normal anesthesia procedures will then be resumed
  The BVGA enables the direct connection of a bag valve device to a Guedel, eliminating the need for a face mask during ventilation The Mask is a classic face mask
  Interventions: Device: Begin with Face-mask

INTERVENTIONS:
Device: Begin with BVGA — Device: BVGA The BVGA enables the direct connection of a bag valve device to a Guedel, eliminating the need for a face mask during ventilation
  Other Names:
  • Bag Valve Guedel Adaptor Device: Face Mask Classic face mask
  Arms: Begin with BVGA
Device: Begin with Face-mask — Device: BVGA The BVGA enables the direct connection of a bag valve device to a Guedel, eliminating the need for a face mask during ventilation
  Other Names:
  • Bag Valve Guedel Adaptor Device: Face Mask Classic face mask
  Arms: Begin with Face-mask

SUMMARY:
Ventilation of a bearded patient with the commonly used face mask has low efficiency because of difficulties to achieve a tight seal around the mouth and nose. The purpose of this study is to evaluate the efficacy of a novel bag valve Guedel adaptor (BVGA) that enables the direct connection of a bag valve device to a Guedel - eliminating the need for a face mask in anesthetized bearded men.

DETAILED DESCRIPTION:
Ventilating a patient using a bag valve and a face mask is not easy to perform, especially for a long period of time, and mandates experience and strength by the care giver. The need for a tight seal around the mouth and nose is a major challenge especially if the patient has a beard. Nevertheless, the face mask is the only approved respiratory support that medics and other basic care givers are allowed to use in the out-of-the-hospital setting, and only physicians and paramedics are allowed to use more advanced techniques, providing a definite airway. Thus, despite its lower effectiveness, the bag valve mask technique is the most commonly used in the field. We have shown previously that the BVGA provides significantly more efficient (less leak) ventilation compared to a facemask, in a randomized, cross-over (BVGA vs mask) controlled clinical trial (NCT02768246) with healthy bearded volunteers that were awake and breathed spontaneously.

The purpose of this study is to evaluate the safety and efficacy of the BVGA compared to a classic facemask in anesthetized bearded volunteers.

Study Design:

Prospective, randomized (sequence randomization), controlled (cross over). The study population will include ASA 1 or 2patients that are planned to undergo elective surgery under general anesthesia with non-depolarizing muscle relaxants. These will include 45 men with beards, and 14 men without beards or women

All subjects will sign an informed consent before participation and will be randomized by sequence (BVGA followed by Mask or Mask followed by BVGA). The physician will initiate anesthesia induction with a face mask according to normal procedures. Experimental phase: According to the sequence of devices determined in the randomization, the physician will then place the first device for 2 minutes, and then replace it with the second device for 2 minutes. The devices will be connected to the operating ventilation machines and physiological and respiratory parameters will be monitored continuously. During the experimental phase, a study assistant will note if the physician used 1 or 2 hands during the ventilation with the experimental devices (BVGA/mask).

The physician will then continue the anesthesia procedures as planned. The physician will complete a questionnaire related to the use of the BVGA in comparison to the standard mask.

ELIGIBILITY:
Inclusion Criteria:

1. Beards men with different levels of beard fullness, men without beards, or women
2. planned to undergo elective surgery with endotracheal intubation using non-depolarizing neuromuscular blocking agents
3. ASA 1 or 2
4. BMI ≤30

Exclusion Criteria:

1. Pregnant women
2. ASA>2
3. Presence of facial fractures or injuries.
4. Expected to suffer from aspiration and requiring rapid sequence induction
5. Edentulous or unstable teeth
6. Morbid obesity
7. Suspected difficult intubation
8. Suspected difficult ventilation (except of the presence of beard)
9. If an unexpected difficulty in ventilation will arise during induction, patient will be excluded from study.
10. Worker from Hadassah Medical Center

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most volunteers are required to have a beard, therefore most volunteers will be men.
Enrollment: 101 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Tidal Volume | 2 minutes
  Tidal volume will be monitored while the volunteer breathes through the BVGA or the face mask. The second minute of each of the interventions will be used for the data analysis.

SECONDARY OUTCOMES:
End tidal CO2 levels (EtCO2) | 2 minutes
  EtCO2 will be monitored while the volunteer breathes through the BVGA or the face mask. The second minute of each of the interventions will be used for the data analysis.
Ease of use | 30 minutes
  The number of hands (1 or 2) the physician had to use during the ventilation procedure while using each device (mask or BVGA)

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Firman, MD, Principal Investigator — Hadassah Medical Organization; Lilach Gavish, PhD, Study Director — Hebrew University of Jerusalem
Locations (1):
- Haddasah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gavish L, Rittblat M, Gertz SD, Shaylor R, Weissman C, Eisenkraft A. Ventilating the Bearded: A Randomized Crossover Trial Comparing a Novel Bag-Valve-Guedel Adaptor to a Standard Mask. Mil Med. 2020 Aug 14;185(7-8):e1300-e1308. doi: 10.1093/milmed/usz378. PMID 33444455